CLINICAL TRIAL: NCT07122076
Title: A Single-arm, Open-label Clinical Study of GT719 Injection for Moderate to Severe Refractory Autoimmune Diseases
Brief Title: GT719 Injection for Moderate to Severe Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-719-003-030
Record Dates: First submitted 2025-07-29; First posted 2025-08-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT719 Injection treatment group (Experimental): GT719 Injection
  Interventions: Biological: GT719 Injection

INTERVENTIONS:
Biological: GT719 Injection — GT719 Injection

SUMMARY:
This study is a prospective single-arm open-label clinical trial, aims to evaluate the safety, efficacy, and cellular pharmacokinetics of GT719 Injection in patients with moderate to severe refractory autoimmune diseases. A total of 10 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria

1. Voluntarily enrolled in the study, signed an informed consent form, willing and able to comply with the study protocol.
2. Aged 18 to 65 years (inclusive), regardless of gender.
3. The functions of important organs meet the following requirements，excluding those attributable to disease activity:

   1. Bone marrow hematopoietic function needs to meet: Neutrophil count ≥1×10^9/L; Hemoglobin ≥80g/L; Platelets ≥30×10^9/L;
   2. Liver function: ALT≤3×ULN; AST≤3×ULN; TBIL≤1.5×ULN;
   3. Renal function: creatinine clearance (CrCl) ≥30 ml/minute;
   4. Coagulation function: International standardized ratio (INR) ≤1.5×ULN, prothrombin time (PT) ≤1.5×ULN;
   5. Heart function: good hemodynamic stability, with no evidence of moderate or greater pericardial effusion.
4. Women of childbearing age must:

   1. During screening, the test result for serum β-human chorionic gonadotropin (β-hCG) was negative;
   2. Agree to avoid breastfeeding during the study period until at least one year after the infusion of GT719 cell injection or until two consecutive flow cytometry tests show the absence of GT719 cells (whichever occurs later);
   3. Male participants with sexual partners and female participants with potential fertility agree to use highly effective contraceptive methods from screening until at least one year after GT719 cell injection or until two consecutive flow cytometry tests show the absence of GT719 cells (whichever occurs later). Male participants must agree to use condoms during sexual contact with pregnant or fertile women for at least one year after infusion of GT719 cell injection, even after successful vasectomy.

Specific inclusion criteria:

Systemic lupus erythematosus

1. Complies with the classification standards of the 2019 European Union Against Rheumatology/American Society of Rheumatology (EULAR/ACR) SLE;
2. Disease activity score SELENA SLEDAI≥6 with at least one Injima Lupus Assessment Group Index (BILAG-2004) category A (severe presentation) or two Category B (moderate presentation) organ scores, or both; Or disease activity score SELENA SLEDAI score ≥8;
3. Definition of relapse refractory: conventional treatment remains ineffective for more than 6 months or disease activity occurs again after remission. Conventional treatment is defined as the use of glucocorticoids and cyclophosphamide, and any of the following immunomodulators: antimalarials, azathioprine, mortemycophanate, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including rituximab, belimumab and telitacicept.

Inflammatory myopathy

1. Inflammatory myopathy fulfilling the 2017 EULAR/ACR classification criteria (including Dermatomyositis (DM), Polymyositis (PM), Anti-Synthetase Syndrome (ASS), and Necrotizing Myopathy (NM)).
2. Positive myositis antibodies;
3. Muscle involvement with Manual Muscle Testing-8 (MMT-8) score less than 142 and at least two abnormalities found among the following five core measurements (Physician Global Assessment (PhGA), Patient Global Assessment (PtGA), or extramuscular disease activity score ≥ 2; Health Assessment Questionnaire (HAQ) total score ≥ 0.25; muscle enzyme levels ≥ 1.5×ULN; or MMT-8 ≥ 142, but with active interstitial lung disease (HRCT showing ground-glass opacities);
4. Definition of relapsed/refractory: Conventional treatment over 6 months remains ineffective, or disease recurrence after remission. Definition of conventional treatment: the use of glucocorticoids and cyclophosphamide, and any one or more of the following immunomodulatory drugs: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab, etc.
5. Definition of progressive: Rapid progression of interstitial lung disease within a short period.

Note: Meeting either criterion 4 or 5 is sufficient.

Diffuse systemic sclerosis

1. Meet the 2013 ACR classification criteria for systemic sclerosis;
2. Positive antibodies related to systemic sclerosis;
3. Definition of relapse refractory: conventional treatment remains ineffective for more than 6 months or disease activity occurs again after remission. Conventional treatment is defined as the use of glucocorticoids and cyclophosphamide, and any of the following immunomodulators: antimalarials, azathioprine, mortemycophanate, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including rituximab, belimumab and telitacicept
4. Definition of progression: rapid skin progression (mRSS increase >25%); Or progression of lung disease (a 10% reduction in FVC, or a more than 5% reduction in FVC with a 15% reduction in DLCO).

Note: Articles 4 and 5 satisfy one or the other.

Exclusion Criteria:

1. SLE participants:

   1. Drug induced SLE;
   2. Patients with lupus crisis or concomitant diseases who require the use of contraindicated drugs according to the protocol are deemed unsuitable for inclusion by the investigator.
2. IIM participants

   1. Documented inclusion body myositis (IBM), drug-induced PM or DM, tumor associated PM or DM, non-inflammatory myopathy (such as muscular dystrophy);
   2. Uncontrolled extramuscular disease damage related to PM or DM:

   ILD: FVC<55% or requiring oxygen therapy;

   Severe swallowing difficulties, as determined by investigator, increase the risk of patients participating in clinical trials;

   Severe cardiac manifestations (such as congestive heart failure, arrhythmia, conduction abnormalities requiring treatment, or myocardial infarction) have been determined by investigator to increase the risk of patients participating in clinical trials.
3. SSc participants

   1. Moderate to severe pulmonary arterial hypertension (PAH) associated with SSc that cannot be controlled by drug therapy;
   2. Rapid progressive SSc related low gastrointestinal (small and large intestine) involvement (requiring parenteral nutrition); Active dilation of gastric antral blood vessels;
   3. Uncontrolled or rapidly progressing ILD with oxygen saturation (SaO2) <92% (in still indoor air); Or require mechanical respiratory assistance (ventilator) within one year prior to signing the informed consent form.
4. Has a history of severe hypersensitivity reactions or allergies;
5. Contraindications or hypersensitivity reactions to any components of fludarabine, cyclophosphamide, and experimental drugs;
6. Suffering from the following heart diseases:

   1. NYHA Grade III or IV congestive heart failure;
   2. Has experienced a myocardial infarction or undergone coronary artery bypass surgery within the 6 months prior to the screening period;
   3. A clinically significant history of ventricular arrhythmia or unexplained syncope, not caused by vasovagal nerve response or dehydration, or a corrected QT interval (QTc)>480 ms during screening;
   4. History of severe non ischemic cardiomyopathy;
7. Any active malignant tumors or history of malignant tumors within the past 5 years before screening. Excluding the following situations: early-stage tumors that have received curative treatment (in situ or stage I tumors, non ulcerative primary melanoma with a depth of<1 mm and no involvement of lymph nodes), basal cell carcinoma of the skin, squamous cell carcinoma of the skin, cervical in situ cancer, or breast in situ cancer that has received potential curative treatment;
8. Individuals with clinically significant bleeding symptoms or clear bleeding tendencies within the 6 months prior to screening, such as gastrointestinal bleeding, hemorrhagic gastric ulcers, etc; Hereditary or acquired bleeding and thrombophilia tendencies (such as hemophilia, coagulation dysfunction, splenic hyperfunction, etc.); Occurrence of arteriovenous thrombosis events within 6 months prior to screening, such as cerebrovascular disease (including cerebral hemorrhage, cerebral infarction, etc.), deep vein thrombosis, and/or pulmonary embolism;
9. When screening, there may be serious underlying medical conditions, such as:

   1. There is evidence to suggest the presence of uncontrollable viruses, bacteria, fungi, or other infections that require systemic intravenous treatment;
   2. There is clear clinical evidence indicating the presence of dementia or changes in mental state;
   3. Any other history of central nervous system disorders or neurodegenerative diseases, such as epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, mental illness;
10. Any of the following test results is positive:

    1. Positive for human immunodeficiency virus (HIV) antibodies;
    2. Hepatitis B surface antigen (HBsAg) positive; Or if the hepatitis B core antibody (HBcAb) is positive and the hepatitis B virus (HBV) - DNA is higher than the detection limit of the analytical method;
    3. Hepatitis C virus (HCV) antibody positive and HCV RNA above the detection limit of the analytical method;
    4. Syphilis antibody positive (false positive result due to reasons other than the disease);
11. Cytomegalovirus (CMV) (DNA) and Epstein Barr virus (EBV) (DNA) tests positive;
12. Active tuberculosis or latent tuberculosis without proper treatment before screening;
13. Received other clinical trial drugs within 4 weeks prior to the signing of the informed consent form (ICF), or the ICF signing date is within 5 half lives of the drug from the last use of the drug in the previous clinical trial (whichever is longer);
14. Received plasma exchange therapy or immunoadsorption therapy within 4 weeks prior to lymphodepleting chemotherapy;
15. Used drugs targeting B cells, including but not limited to rituximab, belimumab, tacrolizumab, etc., within one week before lymphodepleting chemotherapy;
16. Used tacrolimus, cyclosporine, azathioprine, mycophenolate mofetil, mycophenolate mofetil, methotrexate, etc. within 2 weeks before lymphodepleting chemotherapy;
17. Used neonatal Fc receptor (FcRn) antagonist therapy (such as Efgartigimod) within 3 weeks before lymphodepleting chemotherapy;
18. Within 3 weeks prior to lymphodepleting chemotherapy, complement inhibition therapy (such as Ecuzumab) has been used;
19. Received attenuated live vaccine within 4 weeks before lymphodepleting chemotherapy;
20. Having undergone major surgery within the 8 weeks prior to screening, or planning to undergo surgery during the study period;
21. Medical history of organ transplantation;
22. Previously received CAR-T product therapy targeting any target (excluding GT719 therapy);
23. According to the investigator's judgment, the situations that hinder participants from participating in the entire trial, confound the trial results, or participate in the trial that are not in the best interests of the participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2028-08-21 (Estimated); Study Completion 2028-08-21 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing dose limiting toxicity | 28 days
  Proportion of participants experiencing dose limiting toxicity (DLT) within 28 days after cell infusion
Incidence of treatment-emergent adverse events | 3 months
  Safety assessments are conducted using the NCI-CTCAE version 5.0 standards

SECONDARY OUTCOMES:
Efficacy outcomes for SLE | 14 days,1, 2, 3 and 6 Months post GT719 infusion
  SLE Response index 4(SR-4) response: Min/Max Value: Not specified; a decrease in score indicates improvment, higher scores indicate worse outcome
Efficacy outcomes for Systemic Sclerosis | 14 days,1, 2, 3 and 6 Months post GT719 infusion
  ACR-CRISS score (CRISS score≥0.6 improvment, <0.6 no improvement)
Efficacy outcomes for Inflammatory Myopathy | 14 days,1, 2, 3 and 6 Months post GT719 infusion
  Total lmprovement Score (TlS): Min/Max Value: Not specified; an increase in score indicates improvement, higher scores indicate better outcome.

OTHER OUTCOMES:
Efficacy outcomes for SLE | 12 weeks
  SLE Response index 4(SR-4) response: Min/Max Value: Not specified; a decrease in score indicates improvment, higher scores indicate worse outcome
Efficacy outcomes for Systemic Sclerosis | 12 weeks
  ACR-CRISS score (CRISS score≥0.6 improvment, <0.6 no improvement)
Efficacy outcomes for Inflammatory Myopathy | 12 weeks
  Total lmprovement Score (TlS): Min/Max Value: Not specified; an increase in score indicates improvement, higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No